CLINICAL TRIAL: NCT01818648
Title: Acute Effects of a Glucagon-like Peptide 1 Analog, Exenatide, on Gastrointestinal Motor Function and Permeability in Patients With Short Bowel Syndrome on Home Parenteral Nutrition
Brief Title: Exenatide on GI Motor Function and Permeability in Short Bowel Syndrome
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was withdrawn by PI due to decision to study a different medication.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael Camilleri, Primary Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-008505
Record Dates: First submitted 2013-02-28; First posted 2013-03-26 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide (Experimental): Qualifying participants will be assigned to 2 different treatment arms consisting of placebo or exenatide 5 mcg administered subcutaneously twice: the first dose during fasting and the second four hours later. Subsequently, participants will switch over to the alternate treatment arm. In both arms participants will undergo a series of measurements including 24 hour GI transit, permeability measurements by using mannitol and lactulose, and 24 hour urine and stool collections.
  Interventions: Drug: Exenatide
- Placebo (Placebo Comparator): Qualifying participants will be assigned to 2 different treatment arms consisting of placebo or exenatide 5 mcg administered subcutaneously twice: the first dose during fasting and the second four hours later. Subsequently, participants will switch over to the alternate treatment arm. In both arms participants will undergo a series of measurements including 24 hour GI transit, permeability measurements by using mannitol and lactulose, and 24 hour urine and stool collections.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Exenatide — Qualifying participants will be assigned to 2 different treatment arms consisting of placebo or exenatide 5 mcg administered subcutaneously twice: the first dose during fasting and the second four hours later. Subsequently, participants will switch over to the alternate treatment arm. In both arms participants will undergo a series of measurements including 24 hour GI transit, permeability measurements by using mannitol and lactulose, and 24 hour urine and stool collections.
  Arms: Exenatide
Drug: Placebo — Qualifying participants will be assigned to 2 different treatment arms consisting of placebo or exenatide 5 mcg administered subcutaneously twice: the first dose during fasting and the second four hours later. Subsequently, participants will switch over to the alternate treatment arm. In both arms participants will undergo a series of measurements including 24 hour GI transit, permeability measurements by using mannitol and lactulose, and 24 hour urine and stool collections.
  Arms: Placebo

SUMMARY:
We plan to examine the gastrointestinal (GI) physiologic profile of Exenatide, a glucagon-like peptide (GLP-1) analog as a possible intestino-trophic growth factor capable of inducing small bowel adaptation and regeneration in patients with short bowel syndrome (SBS), with the potential to decrease parenteral nutrition dependence.

ELIGIBILITY:
Patients with short bowel syndrome, between the ages of 18-85 who are dependent on parenteral nutrition for at least a year and are being closely followed by the Mayo Clinic Home Parenteral Nutrition Program (HPN) with at least one multisystem evaluation a year.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in 24hr Gastrointestinal and Colonic Transit before and after Exenatide vs placebo | In both arms participants will undergo GI transit measurements on 2 seperate occasions for a total of 24 hours, with a wash out period of 48 hours in between transit studies.
  To measure gastric, small intestinal and colonic (if applicable) transit in patients with short bowel syndrome (SBS) before and after the administration of Exenatide compared to placebo

SECONDARY OUTCOMES:
Change in 24hr Intestinal Permeability before and after administration of Exenatide vs placebo | In both arms participants will undergo intestinal permeability measurements on 2 seperate occasions for 24 hours,with a wash out period of 48 hours in between permeability studies. .
  To measure intestinal permeability to mannitol and lactulose in patients with short bowel syndrome before and after administration of Exenatide compared to placebo

OTHER OUTCOMES:
Change in 24hr Stool Weight before and after administration of Exenatide vs placebo | In both arms participants will collect stool weight for 24 hours in 2 seperate occasions with a wash out period of 48 hours in between collections.
  To measure stool weight in patients with short bowel syndrome before and after administration of Exenatide compared to placebo.
Change in 24hr Urine Volume before and after administration of Exenatide vs placebo | In both arms participants will collect urine volume for 24 hours in 2 seperate occasions with a wash out period of 48 hours in between collections.
  To measure urine volume in patients with short bowel syndrome before and after administration of Exenatide compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic